CLINICAL TRIAL: NCT03433495
Title: Adaptation of Melodic Intonation Therapy to Spanish: a Feasibility and Validation Pilot Clinical Trial
Brief Title: Adaptation of Melodic Intonation Therapy to Spanish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PI-894
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Post Stroke Aphasia
Keywords: stroke; aphasia; melodic intonation therapy
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A neuropsychologist blinded to the patients' clinical characteristics and the group to whom the patient was allocated evaluated outcome variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melodic Intonation Therapy (Active Comparator): The duration of therapy was 12 sessions performed over a 6-week period. Each session lasted 30 minutes. They were performed individually by a speech-experienced therapist previously trained in Melodic Intonation Therapy.
  Interventions: Other: Melodic Intonation Therapy
- Waiting list (No Intervention): No intervention

INTERVENTIONS:
Other: Melodic Intonation Therapy
  Arms: Melodic Intonation Therapy

SUMMARY:
This study was conducted in three phases:

The first phase involved creation of a Spanish adaptation of the Melodic Intonation therapy; the second phase consisted of a pilot non-randomized intervention study to analyse its feasibility for use with 4 Spanish patients with poststroke nonfluent aphasia; the third phase consisted of a pilot randomised, crossover, intervention pilot trial in a different set of patients with poststroke nonfluent aphasia (N=20)

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with nonfluent aphasia due to unilateral stroke in the left hemisphere without neuroimaging evidence of lesions in the right hemisphere who fulfilled the following criteria:

* The time elapsed since the stroke exceeded 6 months.
* Patient had received a standard program of conventional speech therapy after stroke.
* Persistent nonfluent aphasia with the following characteristics:

  * Severely restricted language, which might be limited to meaningless stereotypy; unlike that observed in verbal tasks, the patient might produce some real and relevant words when singing familiar songs.
  * Poor repetition, even for single words.
  * Moderately preserved language comprehension.
  * The nonstereotyped language was produced with a slurring of speech.
  * The total score for the repetition did not exceed the 70th percentile in the Boston Diagnostic Aphasia Examination. The score was obtained from the average score in three areas: repetition of words and repetition of phrases; listening comprehension exceeding the 15th percentile of Boston Diagnostic Aphasia Examination; and from the average score obtained in three areas: word comprehension, commands and complex ideational material.
* The patient was motivated, emotionally stable and had good attention.
* Signed informed consent was provided.

Exclusion Criteria:

* patients with a history of a previous stroke other than the index event or with any clinical condition (e.g., short life expectancy, coexisting disease) or other characteristics that precluded appropriate follow-up in the study
* patients participating in any therapeutic intervention clinical trials evaluating poststroke recovery
* use of psychotropic drugs that interfere with patient evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Communicative Activity Log questionnaire | 6 weeks after the end of therapy
Boston Diagnostic Aphasia Examination | 6 weeks after the end of therapy

IPD SHARING:
Plan to Share IPD: No